CLINICAL TRIAL: NCT01905046
Title: Testing for Atypia in Random Periareolar Fine Needle Aspiration (RPFNA) Cytology After 12 Months Metformin (1, 1-Dimethylbiguanide Hydrochloride) Chemoprevention Versus Placebo Control in Premenopausal Women
Brief Title: Metformin Hydrochloride in Preventing Breast Cancer in Patients With Atypical Hyperplasia or In Situ Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: A211102; U10CA031946 (NIH); NCI-2013-00995 (Registry Identifier: Clinical Trial Reporting Program)
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Atypical Ductal Breast Hyperplasia; BRCA1 Mutation Carrier; BRCA2 Mutation Carrier; Ductal Breast Carcinoma in Situ; Lobular Breast Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: metformin hydrochloride (Experimental): Patients receive metformin hydrochloride PO QD or BID for 24 months. Patients will continue metformin 850 mg PO BID for months 13-24. Patients will undergo RPFNA at 24 months. Follow up visits will be performed at 36 and 48 months after the start of treatment.
  Interventions: Drug: metformin hydrochloride
- Arm II: placebo (Placebo Comparator): Patients receive placebo PO QD or BID for 12 months. Patients may crossover to Arm I for months 13-24.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: metformin hydrochloride — given PO
  Other Names: 1,1 - dimethylbiguanide hydrochloride; 657-24-9; N, N - dimethylimidodicarbonimidic diamide monohydrochloride
  Arms: Arm I: metformin hydrochloride
Other: placebo — given PO
  Other Names: PLCB
  Arms: Arm II: placebo

SUMMARY:
This randomized phase III trial studies metformin hydrochloride to see how well it works compared to placebo in preventing breast cancer in patients with atypical hyperplasia or in situ breast cancer. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of metformin hydrochloride may prevent breast cancer.

DETAILED DESCRIPTION:
I. Test for the presence or absence of cytological atypia (as measured by a Masood Cytology Index Score of 14-17) in unilateral or bilateral random periareolar fine needle aspiration (RPFNA) aspirates after 12 and 24 months (24 month is optional for placebo-only group for patients who remain on placebo arm and will not receive metformin [metformin hydrochloride]) for women receiving metformin versus placebo control. The presence of cytological atypia means any atypia in any RPFNA specimen.

SECONDARY OBJECTIVES:

I. Use the Masood Cytology Index Score to test for the presence of cytological atypia or disappearance of cytological atypia in RPFNA aspirates after 12 months for both arms, and 24 months (24 month is optional for placebo-only group for patients who remain on placebo arm and will not receive metformin, and mandatory for crossover patients) for women receiving metformin 850 mg orally (PO) twice daily (BID) (metformin group).

II. Compare Masood Cytology Score values at 0 and 12 months in right and left breasts (if both breasts were aspirated) from the same individual in the metformin and placebo group.

III. Test the reproducibility of reverse phase protein microarray (RPPM) in duplicate RPPM determinations from individual RPFNA specimens.

IV. Correlate baseline RPPM values with presence of atypia (as measured by Masood Cytology Index Score) at month 12 and month 24 (month 24 optional for placebo-only group; for patients who remain on placebo arm and will not receive metformin) RPFNA.

TERTIARY OBJECTIVES:

I. Test whether metformin alters RPFNA or blood biomarkers associated with breast cancer risk.

II. Test whether metformin alters markers associated with obesity and insulin resistance.

III. Test other exploratory measures in RPFNA and serum including metformin levels and estrogen/progesterone.

IV. Banking: As part of ongoing research for Alliance Cancer Control studies, banking residual blood and RPFNA products for future studies.

ELIGIBILITY:
* PRE-REGISTRATION-INCLUSION CRITERIA
* Must be at increased risk for breast cancer, defined as at least one of the following four criteria:

  * Having had a prior biopsy demonstrating atypical hyperplasia, lobular carcinoma in situ (LCIS), or ductal carcinoma in situ (DCIS)
  * A Gail Model Risk of >= 1.66% over 5 years
  * A strong family history of breast and/or ovarian cancer which is defined as at least one of the following:

    * One first-degree relative with breast cancer before the age of 50 years
    * One first degree relative with bilateral breast cancer
    * Two or more first-degree relatives with breast cancer
    * One first degree relative and two or more second or third degree relatives with breast cancer
    * One first-degree relative with breast cancer and one or more relatives with ovarian cancer
    * Two second or third degree relatives with either breast cancer and one or more with ovarian cancer
    * One second or third degree relative with breast cancer and two or more with ovarian cancer
    * Three or more second or third degree relatives with breast cancer
  * Known breast cancer (BRCA)1 or BRCA2 mutation carrier providing that the woman has

    * Met with a genetic counselor to review genetic testing results, and
    * Has been offered the opportunity to undergo prophylactic mastectomy and oophorectomy
* Pre-menopausal women as defined as four menstrual cycles within the last six months prior to pre-registration; women with less than 4 menses within 6 months prior to pre-registration, or women who have had a hysterectomy with ovaries intact will be considered premenopausal if follicle-stimulating hormone (FSH) level is < 20; women who are using hormonal contraceptives that cause amenorrhea (e.g. injectable and extended oral contraceptives, hormone containing contraceptive ring, or hormone containing intrauterine device) will be considered eligible if they had a minimum of 4 menstrual cycles within the last six months prior to starting on the contraceptive
* Digital mammogram within 365 days prior to pre-registration
* Mammograms must be read as not suspicious for breast cancer (American College of Rheumatology [ACR] class I-III); subjects with a class IV mammogram may be enrolled once they have been evaluated by a breast surgeon and there is no evidence of invasive malignancy
* Must be non-pregnant and non-lactating for at least one year prior to pre-registration
* If currently menstruating, subjects must use a reliable method of birth control
* Willing to provide RPFNA and blood samples for correlative research purposes
* REGISTRATION/RANDOMIZATION INCLUSION CRITERIA:
* Qualifying cytological atypia in RPFNA, Masood score of 14-17; the qualifying RPFNA (of one or both breasts) must be send to Dr. Seewaldt's laboratory for cytological scoring and proteomic analysis; score results must be received from Dr. Seewaldt's lab prior to patient registration/randomization; test must be done =< 90 days prior to registration/randomization

  * Note: Only the contralateral breast can be aspirated in women with DCIS and those undergoing surgery for an atypical lesion; the decision to aspirate the contralateral breast is at the discretion of the woman's surgeon
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 75,000/mm^3
* Creatinine =< 1.4 mg/dL
* Total bilirubin =< 3.0 mg/dL
* Aspartate transaminase (AST) =< 3 x upper limit of normal (ULN)
* Alanine transaminase (ALT) =< 3 x ULN
* Negative pregnancy test done =< 7 days prior to registration/randomization, for women of childbearing potential only

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Women eligible to take tamoxifen must be offered tamoxifen prevention as part of their clinical care and have refused tamoxifen treatment

Exclusion Criteria

* Other active malignancy =< 5 years prior to pre-registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment, i.e., other hormonal therapy, for their cancer
* Body mass index (BMI) < 25
* Receiving Warfarin
* Bilateral breast implants or autologous breast flap reconstruction
* Active diagnosis of alcoholism
* Contraindication to metformin prevention such as acute hypersensitivity or allergic reaction to metformin
* Currently receiving tamoxifen or raloxifene
* Administration of any investigational agent =< 30 days prior to pre-registration
* Previous radiation to both breasts
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving pyrimethamine, cimetidine, rifampin or cephalexin
* Women who have a core biopsy or excisional biopsy containing invasive cancer
* Women who have taken metformin within the past 90 days
* Patients with hemoglobin a1c > 6.3 or who are being actively treated for diabetes

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2025-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Seewaldt, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (27):
- United States (27):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - City of Hope South Pasadena, South Pasadena, California
  - The Community Hospital, Munster, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - M D Anderson Cancer Center, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients receive metformin hydrochloride 850 mg p.o. daily for 4 weeks, then 850 mg p.o. b.i.d. for months 2-12
- Arm II: Patients receive placebo 850 mg p.o. daily for 4 weeks, then 850 mg p.o. b.i.d. for months 2-12. Then patients receive Metformin 850 mg p.o. daily for 4 weeks, then 850 mg p.o. b.i.d. for months 14-24.
Period: Months 0-12
Arm/Group | Arm I | Arm II
Started | 42 | 44
Completed | 42 | 44
Not Completed | 0 | 0
Period: Months 13-24
Arm/Group | Arm I | Arm II
Started | 42 | 44
Completed | 25 | 29
Not Completed | 17 | 15
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 3 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm II: Patients receive placebo 850 mg p.o. daily for 4 weeks, then 850 mg p.o. b.i.d. for months 2-12. Then Metformin 850 mg p.o. daily for 4 weeks, then 850 mg p.o. b.i.d. for months 14-24.
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (6.2) | 41.9 (7.3) | 41.3 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 86
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 35 | 38 | 73
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 37 | 41 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Test for the Presence or Absence of Cytological Atypia in Unilateral or Bilateral RPFNA Aspirates After 12 Months.
Description: Presence of atypia at 12 months is determined through the average of Masood scores across all evaluable breasts for a patient. If the average score is at least 13.5, then patient will be labeled as having atypia. The primary aim of this study is to compare the presence of atypia at month 12 between two arms using the chi-square test in univariable analysis and regressed on group indicator, age, race, stratification factors, and baseline Masood score using logistic regression in multivariable analysis.
Time Frame: 12 months
Population: Per protocol, evaluable patients are defined as having a baseline Masood score between 14 and 17 in at least one breast, and all evaluable breasts undergo satisfactory RPFNA at 12 months. At the time of the primary analysis, we had 66 evaluable patients out of 86 randomized patients (32 Placebo, 34 Metformin).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 32 | 34
Participants
  With Aytpia | 20 | 21
  Without Aytpia | 12 | 13
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p = 0.951, Chi-squared; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.36 to 2.62]

2. Secondary Outcome: Test for the Masood Score and the Presence of Atypia or Disapperance of Atypia in RPFNA After 12 Months (for Both Arms) and 24 Months for Metformin Arm.
Time Frame: Up to 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Compare Masood Cytology Score Value at 0 and 12 in Right and Left Breast From the Same Individual in the Metformin and Non-metformin Group.
Time Frame: Up to 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Test the Reproducibility of RPPM in Duplicate RPPM Determinations From Individual RPFNA Specimens.
Time Frame: Up to 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Correlate Baseline RPPM Values With Presence of Atypia at Month 12 and Month 24.
Time Frame: Up to 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- Arm II Months 0-12: Placebo: Patients receive placebo 850 mg p.o. daily for 4 weeks, then 850 mg p.o. b.i.d. for months 2-12.
- Arm II Months 13-24: Metformin: Patients recieve metformin 850 mg p.o. daily for 4 weeks, then 850 mg p.o. b.i.d. for months 14-24.
Arm/Group | Arm I | Arm II Months 0-12: Placebo | Arm II Months 13-24: Metformin
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/44 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/44 | 2/57
Other Adverse Events (participants affected / at risk) | 24/42 | 34/44 | 32/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=42) | Arm II Months 0-12: Placebo (N=44) | Arm II Months 13-24: Metformin (N=57)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=42) | Arm II Months 0-12: Placebo (N=44) | Arm II Months 13-24: Metformin (N=57)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (3)
Bloating (Gastrointestinal disorders) | 6 (7) | 12 (17) | 10 (11)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 12 (19) | 26 (35) | 24 (34)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (4) | 2 (2) | 4 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 14 (21) | 14 (19)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 8 (9) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2) | 3 (3)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (3) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT01905046/Prot_SAP_000.pdf